CLINICAL TRIAL: NCT01573819
Title: A Randomised, Placebo Controlled, Ascending, Repeat Dose Study in Healthy Volunteers Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK356278
Brief Title: A Repeat Dose Study in Healthy Volunteers Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK356278
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 115719
Record Dates: First submitted 2012-02-16; First posted 2012-04-10 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Huntington Disease
Keywords: repeat dose; PDE4; healthy volunteers; GSK356278
MeSH Terms: conditions — Huntington Disease | interventions — 5-(5-((2,4-dimethylthiazol-5-yl)methyl)-1,3,4-oxadiazol-2-yl)-1-ethyl-N-(tetrahydro-2H-pyran-4-yl)-1H-pyrazolo(3,4-b)pyridin-4-amine

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Cohort 1 (Experimental): A dose of 2mg per day for 10 days
  Interventions: Drug: GSK356278; Drug: Placebo
- Cohort 2 (Experimental): A dose of Xmg for 14 days. the dose will be determined from Cohort 1 not to exceed 14 mg
  Interventions: Drug: GSK356278; Drug: Placebo
- Cohort 3 (Experimental): a single dose of Ymg with a wash out of 7 days followed by 28 days of repeat dosing. The dose (Ymg) will be determined from cohort 1 and 2 not to exceed 14 mg.
  Interventions: Drug: GSK356278; Drug: Placebo

INTERVENTIONS:
Drug: GSK356278 — Cohort 1: A dose of 2mg per day for 10 days; Cohort 2: A dose of Xmg for 14 days. the dose will be determined from Cohort 1 not to exceed 14 mg; Cohort 3: a single dose of Ymg with a wash out of 7 days followed by 28 days of repeat dosing. The dose (Ymg) will be determined from cohort 1 and 2 not to exceed 14 mg.
Drug: Placebo — Cohort 1, a placebo per day for 10 days Cohort 2, a placebo per day for 14 days Cohort 3, a single placebo with a wash out of 7 days followed by 28 days of repeat dosing of a placebo per day.

SUMMARY:
The study drug, GSK356278, is a possible new medicine for the treatment of Huntington's disease. Huntington's disease, which is often called HD, is caused by a faulty gene that is passed down through families. HD causes damage to nerve cells in the brain which causes them to waste away. As the damage progresses patients develop symptoms that affect every aspect of life. HD reduces people's ability to walk, talk, think, communicate and causes uncontrolled movements. GSK356278 may slow down the progression of damage to nerve cells in people with HD and help with their ability to think.

GSK356278 was well tolerated when it was given as a single dose to healthy people. In this study we want to see what effects, both good and bad, GSK356278 has in people when it is taken every day. During the study we will look at about 3 different doses of GSK356278 in about 36 healthy people. The study will also look at how GSK356278 tablets behave in the body after it is swallowed (this is called pharmacokinetics). The study will also look at effects of GSK356278 on the body (this is called pharmacodynamics). The study will help to design future clinical studies with GSK356278.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than and equal to 1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinically significant abnormality or laboratory parameters significantly outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential is defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) greater than 40 MlU/ml and estradiol less than 40 pg/ml (less than 147 pmol/L) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will not be eligible for the study.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol (contraception requirements). This criterion must be followed from the time of the first dose of study medication until the follow up visit.
* Body weight greater than and equal to 50 kg and BMI within the range 19 - 30 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.Average of triplicate QTcF less than 450 msec (on an average of triplicate values)
* Normal echocardiography, plasma troponin and BNP levels confirmed before first dose

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of greater than 21 units for males or greater than 14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 ml) of beer, 1 glass (125ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 30 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco or nicotine-containing products within 6 months prior to screening.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids from 7 daysprior to the first dose of study medication.
* Any history of suicidal behaviours or any suicidal ideation of type 4 or 5 on the CSSR in the last six months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-11-24 (Actual); Primary Completion 2012-04-02 (Actual); Study Completion 2012-04-02 (Actual)

PRIMARY OUTCOMES:
Composite (or Profile) of Pharmacokinetics | Cohort 1 for 288 hours post dose; Cohort 2 for 384 hours post dose; Cohort 3 single dose session for 72 hours; Cohort 3 repeat dose session for 744 hours post dose.
  The primary pharmacokinetic endpoints following oral administration are: peak plasma concentration (Cmax), time of peak plasma concentration (tmax), area under the plasma concentration-time curve over the dose interval , and area under the plasma concentration-time curve from time-zero extrapolated to infinite time, accumulation ratio (Ro), terminal half-life (t½ ), apparent oral clearance (CL/F) and trough concentration.
Safety and tolerability parameters including change from baseline measures for vital signs | Cohort 1 for 15 days post dose; Cohort 2 for 19 days post dose; Cohort 3 single dose session for 4 days post dose; Cohort 3 repeat dose for 33 days post dose.
Safety and tolerability parameters including change from baseline for 12-lead ECGs | Cohort 1 for 15 days post dose; Cohort 2 for 19 days post dose; Cohort 3 single dose session for 4 days post dose; Cohort 3 repeat dose for 33 days post dose.
Safety and tolerability parameters including change from baseline for telemetry ECGs | Cohort 1 for 8 hours 30 minutes on Day 1 and Day 10; Cohort 2 for 8 hours 30 minutes on Day 1 and Day 14; Cohort 3 single dose session for 8 hours 30 minutes on Day 1; Cohort 3 repeat dose for 8 hours 30 minutes on Day 1 on Day28.
Safety and tolerability parameters including change from baseline for clinical laboratory tests | Cohort 1 for up to 28 days; Cohort 2 for up to 32 days; Cohort 3 single dose for 2 days; Cohort 3 repeat dose for up to 46 days
  hematology, chemistry, liver function enzymes, troponin, B-type natriuretic peptide, inflammatory markers (Haptoglobin, fibrinogen, CRP, IL-6) and urinalysis
Safety and tolerability parameters including change from baseline for clinical lab tests | Cohort 1 for 11 days; Cohort 2 for 15 days; Cohort 3 single dose for 2 days; Cohort 3 repeat dose for 29 days
  Inflammatory markers (Haptoglobin, fibrinogen, CRP, IL-6)
Safety and tolerability parameters including change from baseline for echocardiography | Cohort 1 for 12 days; Cohort 2 for 16 days; Cohort 3 repeat dose for 30 days
Safety and tolerability parameters including change from baseline for Bond and Lader VAS | Cohort 1 for 10 days; Cohort 2 for 14 days; Cohort 3 single dose for 2-3 hours post dose on Day 1; Cohort 3 repeat dose for 28 days
Safety and tolerability parameters including change from baseline for Columbia Suicide Severity Rating Scale (C-SSRS) | Cohort 1 for 14 days; Cohort 2 for 18 days; Cohort 3 repeat dose for 32 days
Safety and tolerability parameters including change from baseline for Rhodes Index of Nausea, Vomiting and Retching | Cohort 1 for 11 days; Cohort 2 for 15 days; Cohort 3 single dose for 2 days; Cohort 3 repeat dose for 28 days
Safety and tolerability parameters including change from baseline in the collection of adverse events | Cohort 1 for 14 days; Cohort 2 for up to 32 days; Cohort 3 single dose for 4 days; Cohort 3 repeat dose for up to 46 days

SECONDARY OUTCOMES:
Pharmacodynamic parameters including change from baseline for electroencephalography | Cohort 2 for 13 days Cohort 3 repeat dose for 25 days
Pharmacodynamic parameters including change from baseline for cognition test | Cohort 2 for 12 days Cohort 3 repeat dose for 26 days
Pharmacodynamic parameters including change from baseline for plasma Brain-derived neurotrophic factor | Cohort 1 for 11 days; Cohort 2 for 15 days; Cohort 3 single dose session for 2 days; Cohort 3 repeat dose session for 29 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Zuidlaren, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115719 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115719?search=study&search_terms=115719#rs
- Available data/document: Annotated Case Report Form: 115719 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115719 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115719 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115719 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115719 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115719 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115719 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register